CLINICAL TRIAL: NCT01824212
Title: Recognizing Ventricular Fibrillation From an Area of a Mobile Phone
Status: Completed | Type: Observational
Sponsor: North Karelia Central Hospital (Other)
Collaborators: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Sakari Syvaoja, MD, North Karelia Central Hospital
Other Study IDs: NKCHAne001
Record Dates: First submitted 2013-03-27; First posted 2013-04-04 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Ventricular Fibrillation
Keywords: Ventricular fibrillation; Cardiac arrest; Mobile technology
MeSH Terms: conditions — Ventricular Fibrillation; Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICD-patients: Patients to whom cardiac fibrillation will be induced during the implantation of an implantable cardioverter defibrillator (ICD) or patients with an already implanted ICD, which function needs to be revised and during the revision cardiac defibrillation will be induced.

SUMMARY:
Recognition of out of hospital cardiac arrest (OHCA) during an emergency call is based on standardized questions concerning the symptoms of OHCA. With this method cardiac arrest is recognized in 50-83% of cases. When the emergency medical dispatcher identifies cardiac arrest during the emergency call the survival of the patient improves. Accurate emergency medical service response is activated promptly and bystander will receive cardiopulmonary resuscitation (CPR) instructions. It has been estimated that proper implementation of CPR instructions will save thousands of lives each year.

If the ECG could be recorded by the mobile phone, transmitted during the emergency call to the dispatch centre and analysed there with the software of a semi-automated external defibrillator(AED), the recognition of cardiac arrest could be more accurate.

The aim of this study is to examine, if AED, with minimal size electrodes within an area of a mobile phone, is able to recognize reliably ventricular fibrillation (VF), the rhythm with the best prognosis in OHCA.

DETAILED DESCRIPTION:
Dysrhythmia patients who need an implantable cardioverter defibrillator(ICD) or patients with an already implanted ICD which function needs to be revised will be recruited into this study. Our hypothesis is that the ECG and VF is recordable in 100% of cases with a semi-automatic defibrillator. In sample size calculations we compared this 100% recognition to the present situation with 80% recognition of cardiac arrest in emergency medical communication centre during emergency call. According to the power calculation of 1-sided binomial test with risk level 0.05 and power of 95 %, 22 observations is needed to detect difference between expected full successes (99 %) from the previous 80 % of successes in recognition.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* ventricular fibrillation will be induced during the implantation or revision of ICD
* patient's informed consent

Exclusion Criteria:

* ventricular fibrillation will not be induced during the implantation or revision of ICD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe dysrhytmia and the necessity to an implantable cardioverter defibrillator (ICD)
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2013-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The ability of AED to recognise induced VF | 24 hours
  The ability of AED to correctly recognise ventricular fibrillation from a bipolar ECG recorded within an area of mobile phone: is the recognition good enough to automatically divide the rhythm correctly into categories of shockable and non-shockable?

SECONDARY OUTCOMES:
Quality of VF | 24 hour
  The recorded rhythms will be analysed, beside an AED, by two experienced cardiologists and categorised as shockable or non-shockable. The cardiologists also will assess the quality of the recordings and grade each recording according to three categories of quality: 1, bad; 2, average; 3, good.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Jäntti, MD, PhD, Study Director — Kuopio University Hospital; Sakari Syväoja, MD, Principal Investigator — North Karelia Central Hospital
Locations (2):
- Finland (2):
  - North Karelia Central Hospital, Joensuu
  - Kuopio University Hospital, Kuopio